CLINICAL TRIAL: NCT01657149
Title: Influence of Manual Lymph Drainage During Hospitalization on Swelling, Function and Pain in Patients After Total Knee Replacement - Randomized Control Trial.
Brief Title: Influence of Manual Lymph Drainage During Hospitalization on Swelling, Function and Pain in Patients After Total Knee Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: a cardinal member of The research team withdrawn from study, the study has beem terminated.
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0081-12-RMC
Record Dates: First submitted 2012-07-15; First posted 2012-08-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2015-08

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Research Group (Experimental): receive lymphatic massage and individual physiotherapy
  Interventions: Procedure: Lymphatic massage and individual physiotherapy
- Control group (Active Comparator): receive individual physiotherapy only
  Interventions: Procedure: individual physiotherapy only

INTERVENTIONS:
Procedure: Lymphatic massage and individual physiotherapy — lymphatic massage and individual physiotherapy
  Arms: Research Group
Procedure: individual physiotherapy only — individual physiotherapy only
  Arms: Control group

SUMMARY:
To investigate the effects of lymphatic drainage massage performed immediately after total knee replacement in relation to reduction of limb circumference, pain reduction and functional improvement.

DETAILED DESCRIPTION:
In the past few decades there has been a rise in the number of knee replacements performed due to degenerative arthritis. In general over the years the number of operations has risen while the age of the patients has gone down. The aim of these operations is to improve quality of life, alleviate pain and improve function.

Post operative complications can delay recovery and rehabilitation, lengthen hospitalization duration and in extreme cases lead to failure of the operation. These complications include infection, deep vein thrombosis, swelling and edema, pain, impairment of range of motion, muscle weakness and functional disability.

Reduction of post operative edema may help to speed up recovery after total knee replacement.

Recently an effective treatment has been found for lymphatic edema that appears after oncological operations that include removal of lymph nodes or due to blood vessel disorders. This treatment is administered by a physiotherapist and includes lymphatic drainage massage, compression bandaging and exercises.

This trial will examine the effect of lymphatic massage treatment on orthopedic patients to ascertain if the use of this technique can shorten the duration and improve the quality of the post operative rehabilitation and prevent other post operative complications. At the present time not enough research has been done in this field and it is necessary to continue to investigate the efficiency of the lymphatic treatment in acute orthopedic patients.

Aims To investigate the effects of lymphatic drainage massage performed immediately after total knee replacement in relation to reduction of limb circumference, pain reduction and functional improvement.

Methods This blind randomized trial will take place in the Sharon hospital in Petach Tikvah with the cooperation of the orthopedic surgeons. The patients will be randomized into two groups- each containing 15 patients. The research group will receive lymphatic massage and individual physiotherapy while the control group will receive individual physiotherapy only.

Methods In order to assess the effects of the treatment the primary measurement will be circumferential measurement of limb volume. The secondary measurements will be pain assessment according to the VAS scale, a functional assessment according to BI"TI and range of motion measured with an inclinometer .

The measurements will be taken once prior to hospitalization. During hospitalization the measurements will be taken daily including the day of the release home and one last measurement will be taken 6 weeks after the operation. All measurements are valid and reliable.

The trial is scheduled to last 3-4 months

ELIGIBILITY:
Inclusion Criteria:

* primary total knee replacement
* ages 50-85
* preserved cognitive facilities and comprehension.

Exclusion Criteria:

* Severe chronic heart failure.
* previous episode of lymph edema.
* surgical removal of lymph nodes in the lower limbs.
* significant scarring of the lower limbs (larger than 10 cm).
* Deterioration in a patient's medical condition or an infection of the lower limb during the trial period will also cause exclusion of that patient.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Circumferential measurement of limb volume | The circumferential measurements will be assesed pre operative and post operative on daily basis for 5 days post op

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) Inclinometer | VAS & INCLINOMETER will be assessed on a daily basis for 5 days post op
Daily functional capacity Assessment | Daily functional capacity Assessment after 6 days post op. All Outcomes will be reassessed after 6 weeks post op

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Campus Golda, Petah Tikva, Israel